CLINICAL TRIAL: NCT06580535
Title: Impact of Estrogen Receptor Modulators on Mania Patients and Its Relationship With Genetic Polymorphism of Phospholipase C Epsilon1
Brief Title: Effect of Esterogen Receptor Modulator on Gene in Bipolar Diseas
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Kamal Fahmy, Demonstrator, Assiut University
Other Study IDs: bipolar disorder
Record Dates: First submitted 2024-05-31; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Bipolar Disorder
Keywords: Mania
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood sample for detection of PLCE1 gene polymorphism in bipolar disorder
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1 (patients): 50 patients assigned to receive treatment of bipolar disorder
  Interventions: Other: blood sample
- Group 2 recrutied blood from patients: GroupII:50 blood sample will be recruited from G1for in vitro tissue culture to study the effect of tamoxifen on the WBCs of patients
  Interventions: Other: blood sample
- group 3 control: GroupIII:50 healthy control will be recruited (age and sex will be matched
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — Blood sample taking from patient for tissue culture

SUMMARY:
1. Identify randomized controlled trials of tamoxifen (Estrogen Receptor modulator) in in addition to traditional treatment of bipolar disorder and synthesize the results using meta-analysis.
2. Systematically estimate the effects of Phospholipase C epsilon 1 gene (PLCE1) rs2274223and gene polymorphism on the susceptibility to treatment.
3. Study the pathway involved in the action of tamoxifen by incorporating TMX into nanoparticles and evaluating tyrosine kinase in responders WBCS culture and evaluate nanoparticle as a hope for future treatment of CNS disorders.

DETAILED DESCRIPTION:
Bipolar disorder, formerly known as manic depression, is typified by severe mood fluctuations with emotional highs (mania or hypomania) and lows (depression). Tamoxifen [TMX], an oral medication, has been proposed as a potential treatment for bipolar disorder. Tamoxifen)modulator of the Estrogen Recptor) functions by blocking the intracellular action of protein kinase C, which is the mechanism by which popular treatments for bipolar disorder such as valproate and lithium function. . Targeted therapy benefits greatly from drug delivery methods based on nanoparticles because they enhance bioavailability, decrease side effects, and increase efficiency. .

Enzymes belonging to the PKC class are essential for cell signaling. Data from previous studies suggest that increased PKC activity may affect the prefrontal cortical regulation of behavior and thinking. PKC is unique in that it is controlled by tyrosine phosphorylation and has several subcellular destinations . In a study of bipolar individuals who responded well to lithium, a variant in the phospholipase C gene, which codes for the first enzyme in the PKC cascade, was discovered .

The 26th exon of the Phospholipase C epsilon1gene (PLCE1) gene contains the non-synonymous SNP Rs2274223, which can change one amino acid from histidine to arginine 6. SNP rs2274223 in PLCE1 is one of the polymorphic loci that has been studied the most .

ELIGIBILITY:
Inclusion Criteria:

1. Fifty subjects 2.15-70 years of age 3.recently diagnosed as bipolar disorder 4.assigned to receive traditional treatment of bipolar disorder

Exclusion Criteria:

1. Patients who have a concurrent sever illness like cancer ,liver disease
2. receiving additional treatment

Ages: 15 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: GroupI:50 patients assigned to receive treatment of bipolar disorder GroupII:50 blood sample will be recruited from G1for in vitro tissue culture to study the effect of tamoxifen on the WBCs of patients GroupIII:50 healthy control will be recruited (age and sex will be matched)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
change in Young Mania Rating Scale(YMRS) Score | e.g.4 weeks
  Mean change in YMRS score from baseline to the end of treatment (range:0-60;higher score indicate sever mania)

SECONDARY OUTCOMES:
Percentage of Participants with Treatment Response | e.g.,4 weeks
  Percentage of participants with a ≥50% reduction in attack rating scores from baseline to end of treatment.

REFERENCES:
- [Background] Kishi T, Ikuta T, Matsuda Y, Sakuma K, Okuya M, Nomura I, Hatano M, Iwata N. Pharmacological treatment for bipolar mania: a systematic review and network meta-analysis of double-blind randomized controlled trials. Mol Psychiatry. 2022 Feb;27(2):1136-1144. doi: 10.1038/s41380-021-01334-4. Epub 2021 Oct 12. PMID 34642461
- [Background] Yetisgin AA, Cetinel S, Zuvin M, Kosar A, Kutlu O. Therapeutic Nanoparticles and Their Targeted Delivery Applications. Molecules. 2020 May 8;25(9):2193. doi: 10.3390/molecules25092193. PMID 32397080
- [Background] Palmer AJ, Lochhead P, Hold GL, Rabkin CS, Chow WH, Lissowska J, Vaughan TL, Berry S, Gammon M, Risch H, El-Omar EM. Genetic variation in C20orf54, PLCE1 and MUC1 and the risk of upper gastrointestinal cancers in Caucasian populations. Eur J Cancer Prev. 2012 Nov;21(6):541-4. doi: 10.1097/CEJ.0b013e3283529b79. PMID 22805490
- [Background] Hu H, Yang J, Sun Y, Yang Y, Qian J, Jin L, Wang M, Bi R, Zhang R, Zhu M, Sun M, Ma H, Wei Q, Jiang G, Zhou X, Chen H. Putatively functional PLCE1 variants and susceptibility to esophageal squamous cell carcinoma (ESCC): a case-control study in eastern Chinese populations. Ann Surg Oncol. 2012 Jul;19(7):2403-10. doi: 10.1245/s10434-011-2160-y. Epub 2011 Dec 28. PMID 22203178
- [Background] Zhang Y, Li W, Wang Y, Wang N. The PLCE1 rs2274223 variant is associated with the risk of laryngeal squamous cell carcinoma. Int J Med Sci. 2020 Oct 8;17(17):2826-2830. doi: 10.7150/ijms.49012. eCollection 2020. PMID 33162810
- [Background] Khan Z, Sattar S, Abubakar M, Arshed MJ, Aslam R, Shah STA, Javed S, Tariq A, Manzoor S, Bostan N. Preparation and in Vitro Evaluation of Tamoxifen-Conjugated, Eco-Friendly, Agar-Based Hybrid Magnetic Nanoparticles for Their Potential Use in Breast Cancer Treatment. ACS Omega. 2023 Jul 14;8(29):25808-25816. doi: 10.1021/acsomega.3c00844. eCollection 2023 Jul 25. PMID 37521645